CLINICAL TRIAL: NCT00641498
Title: Effectiveness of Standard Emergency Department Psychiatric Treatment Compared With Effectiveness of Standard Emergency Department Psychiatric Treatment Associated With Treatment Delivery by a Suicide Prevention Center.
Brief Title: Effectiveness of Standard Emergency Department Psychiatric Treatment Associated With Treatment Delivery by a Suicide Prevention Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0601401; PHRC suicide
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Suicide Attempted
Keywords: suicide; parasuicide; prevention; individual supportive psychotherapy
MeSH Terms: conditions — Suicide, Attempted; Suicide | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Usual therapy
- Active group (Experimental): Individual supportive psychotherapy initiated in the Emergency department
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — Individual supportive
  Arms: Active group

SUMMARY:
Very few studies have proved the effectiveness of treatment for suicide attempt patients. Our objective is to evaluate the addition of the resources of an suicide prevention centre to standard psychiatric treatment in the Emergency Department. Consecutive suicide attempt patients in 2 Emergency departments (multicenter study) were included after standard psychiatric treatment and referral. After Written informed consent, psychological assessment (depression, suicide intention) was carried out After randomisation, control patients were given an information card describing the Suicide Prevention Center (SPC); experimental patients had a first meeting with a psychologist of the SPC.

To verify the hypothesis of a decrease in suicidal behaviors in the experimental group, an evaluation of these behaviors was carried out every month during a two year follow-up.

DETAILED DESCRIPTION:
Very few studies have proved the effectiveness of treatment for suicide attempt patients. Our objective is to evaluate the addition of the resources of an existent suicide prevention centre to standard psychiatric treatment in the Emergency Department. Consecutive suicide attempt (self poisoning) patients in 2 Emergency departments (multicenter study) were included after standard psychiatric treatment and referral. After Written informed consent, psychological assessment (depression, suicide intent scale/SIS Beck Depression Inventory, Toronto Ale, Beck Hopelessness Sc, Audit, mini, PDQ 4) was carried out After randomisation, control patients were given an information card describing the Suicide Prevention Center (SPC); experimental patients had a first meeting with a psychologist of the SPC. The number of subjects included should be 405 per group. To verify the hypothesis of a decrease in suicidal behaviors in the experimental group, an evaluation of these behaviors was carried out every month during a two year follow-up The frequency of subsequent suicidal behavior will be monitored by the scrutiny of the Emergency Dept records. Death by suicide will be identified by the examination of information obtained from the national death statistics office (INSERM).

ELIGIBILITY:
Inclusion Criteria:

* parasuicide by self-poisoning
* Glasgow score=15
* Standard psychiatric treatment

Exclusion Criteria:

* No speaking french
* committed inpatient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2007-03; Primary Completion 2009-12 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Suicide behavior defined by self poisoning or other suicidal attempts in the emergency departments of the region. Death by suicide will be identified by the examination of information obtained from the national death statistics office (INSERM). | 2 years

SECONDARY OUTCOMES:
Level of depression, suicide ideation, level of despair, level of alexithymia | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BIRMES, PhD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - Service d'Accueil des Urgences, Brive-la-Gaillarde
  - Laboratoire de Stress Post-Traumatique, Toulouse

REFERENCES:
- [Derived] Cailhol L, Marcoux M, Mathur A, Yrondi A, Birmes P. Predictors of prospective suicide attempts in a group at risk of personality disorder following self-poisoning. Front Psychiatry. 2023 Jun 9;14:1084730. doi: 10.3389/fpsyt.2023.1084730. eCollection 2023. PMID 37363177
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617